CLINICAL TRIAL: NCT02665988
Title: A Single-Blind, Randomized Control Trial of Adjunctive Transcranial Direct Current Stimulation (tDCS) for Chronic Pain Among Patients Receiving Specialized, Inpatient Multi-Modal Pain Management
Brief Title: Adjunctive Transcranial Direct Current Stimulation
Acronym: tDCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We terminated the study because the Pain Management Program closed in January 2018.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Alok Madan, Director, Pain Management Program at The Menninger Clinic, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-36721
Record Dates: First submitted 2016-01-22; First posted 2016-01-28 (Estimated); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Chronic Pain; Psychiatric Disorders
Keywords: Transcranial Direct Current Stimulation
MeSH Terms: conditions — Chronic Pain; Mental Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real tDCS (Experimental): Those receiving experimental treatment will receive real tDCS during 20-minute periods over the course of 10 sessions. The treatment will be delivered by trained clinical personnel.
  Interventions: Device: tDCS
- Sham tDCS (Placebo Comparator): Those receiving sham tDCS will receive active tDCS during 20-minute periods over the course of 10 sessions. The treatment will be delivered by trained clinical personnel.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: tDCS — Prior to initiating the real tDCS trial and to reduce the likelihood of irritation associated with electrical stimulation, a low dose (1/8 of an inch) topical lidocaine (4%) cream will be applied to the skin where the tDCS the sponge-coated, surface electrodes soaked in saline solution will be placed. Neurotargeting tDCS-explorer software, Version 2.3 will be used to locate the left and right DLPFC, where anodal stimulation of the left DLPFC and cathodal stimulation of the right DLPFC will be received. Real tDCS will be applied during 20-minute periods over the course of 10 sessions. After each session, vitamin-E will be applied to the skin where the electrodes had been placed to reduce likelihood of skin irritation.
  Other Names: transcranial Direct Current Stimulation
  Arms: Real tDCS
Device: Sham tDCS — Participants randomized to sham tDCS will undergo the same procedures as those in the real tDCS sample, including the same pre-treatment lidocaine 4% cream, localization of electrode placement, actual placement of electrodes, turning on the tDCS device in sham setting but will not receive actual stimulation during the 20 minutes of each session, as well as post-treatment vitamin E.
  Other Names: Sham transcranial Direct Current Stimulation
  Arms: Sham tDCS

SUMMARY:
Transcranial direct current stimulation (tDCS) is an investigational device that has not been approved for the treatment of any medical condition by the FDA but is allowed to be used for research purposes. In clinical trials tDCS has been associated with pain relief by decreasing the intensity and duration of chronic pain. tDCS potentially works by stimulating the brain by delivering an extremely low-level electrical current to areas below the forehead - areas associated with chronic pain. It is anticipated that this current will increase brain activity or the likelihood of brain activity in these areas, affecting individual's ability to regulate pain.

The purpose of this study is to compare eligible participants in the Pain Management Program at The Menninger Clinic receiving adjunctive real transcranial Direct Current Stimulation (tDCS) versus those receiving sham tDCS in the resolution of chronic pain. The primary objectives are: (1) improving pain tolerance and (2) improving subjective pain experience. Secondary objectives are: (1) improving subjective experience of sleep quality and (2) increasing physical activity.

DETAILED DESCRIPTION:
Chronic or persistent pain is pain that continues when it should not be present; it is ongoing or recurrent pain, lasting beyond the usual course of acute illness or injury, and which unfavorably affects the individual's well-being. The Institute of Medicine (2011) estimates that 116 million American adults experience chronic pain with direct and indirect costs to the US economy totaling in excess of half a trillion dollars annually. Current treatments for chronic pain are only partially effective, especially when used alone. There is a critical need to develop new and more effective treatments for chronic pain. Transcranial Direct Current Stimulation (tDCS) may be helpful as an additional treatment for patients with chronic pain.

Doctors and scientists conducting this research study want to evaluate the effectiveness of an investigational device (tDCS) that delivers a form of brain stimulation as an additional treatment to standard of care in the Menninger Clinic's Pain Management Program. Stimulation with tDCS as an adjunctive to medication-based treatments as well non-medication treatments options (such as physical therapy and psychotherapy) may improve an individual's ability to tolerate the physical and emotional distress associated with chronic pain. Therefore the investigators propose to engage in a clinical trial of adjunctive tDCS for chronic pain, restricting enrollment to the population receiving services in the Pain Management Program.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females greater than equal to 18 years old.
2. Females with a confirmed negative pregnancy test (which is conducted within 24 hours of admission to the hospital as part of standard of clinical care).
3. Confirmed diagnosis of chronic pain.
4. Must be admitted to the Pain Management Program at The Menninger Clinic.

Exclusion Criteria:

1. Presence of actively psychosis, cognitively impairment.
2. Contraindications to tDCS:

   1. Presence of any preexisting irritation, cuts, or lesions where the tDCS will be placed (i.e., the forehead).
   2. Presence of any preexisting unstable medical conditions, or conditions that may increase the risk of stimulation such as uncontrolled epilepsy.
   3. Presence of history of severe cranial trauma with alteration of the cranial anatomy or metallic intracranial implants.
3. None fluent in the English language.
4. Presence of known sensitivity to Lidocaine 4%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alok Madan, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- The Pain Management Program at The Menninger Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Description of data may affect potential subject's awareness of sham versus real transcranial Direct Current Stimulation (tDCS)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real tDCS | Sham tDCS
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real tDCS | Sham tDCS | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) for Pain Change From Baseline
Description: Visual analogue scale measure for pain. Score range from 0-10. For rating overall pain, ranging from none, mild, moderate, or severe pain.
Time Frame: On a weekly basis: 1) Day 1 (first day of tDCS). 2) Day 8 (after first week with post 5 consecutive sessions of tDCS followed by 2 consecutive days without tDCS). 3) Day 15 (after second week post another 5 sessions of tDCS followed by 2 consecutive days
Population: Analyses were not performed. Given the premature termination of the clinical program, the limited sample size of participants completing the study, the heterogeneity of chronic pain etiology and psychiatric comorbidity among participants, as well as variable and personalized interventions delivered as a part of the clinical care participants received, the data collected would have been grossly underpowered to provide meaningful results.
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants reported adverse events daily during each day of stimulation (prior to the actual stimulation) as well as weekly for two weeks following the active phase of the trial. Data were collected for 22 days during the following days: days 1-5, days 8-12, day 15, and day 22.
Arm/Group | Real tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT02665988/Prot_SAP_000.pdf